CLINICAL TRIAL: NCT03989336
Title: A Randomized, Single-blind, Placebo-controlled, Phase 2 Study to Evaluate the Safety and Efficacy of the Pan-immunotherapy in Subjects With Relapsed/Refractory Ovarian Cancer
Brief Title: A Study of the Pan-immunotherapy in Patients With Relapsed/Refractory Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-040
Record Dates: First submitted 2019-06-15; First posted 2019-06-18 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Ovarian Cancer
Keywords: relapsed; refractory; anti-PD-1 antibody; Manganese; chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — manganese chloride; 130-nm albumin-bound paclitaxel; Paclitaxel; Injections; sintilimab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manganese primed Sintilimab plus nPP chemotherapy (Experimental): Subject received Manganese primed Sintilimab, nab-paclitaxel and platinum chemotherapy every 3 weeks until achieving a second assessable complete response or progressive disease, development of unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Manganese Chloride; Drug: nab-paclitaxel; Drug: Platinum chemotherapy; Drug: Sintilimab
- Sintilimab plus nPP chemotherapy (Active Comparator): Subject received Sintilimab, nab-paclitaxel and platinum chemotherapy every 3 weeks until achieving a second assessable complete response or progressive disease, development of unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: nab-paclitaxel; Drug: Platinum chemotherapy; Drug: Sintilimab

INTERVENTIONS:
Drug: Manganese Chloride — Administered by inhalation at 0.4mg/kg twice per week in the first 3-week cycle, and then inhaled 0.4mg/kg twice in the first week of each 3-week cycle thereafter
  Arms: Manganese primed Sintilimab plus nPP chemotherapy
Drug: nab-paclitaxel — Administered intravenously, 180-220mg/m2 on day 2 in a 3-week cycle (day 1 without Manganese priming)
  Other Names: Paclitaxel For Injection (Albumin Bound)
Drug: Platinum chemotherapy — Administered intravenously, Cisplatin (60-80mg/m2) or Carboplatin (area under the curve [AUC] 4-6 mg/mL per min) on day 2 in a 3-week cycle (day 1 without Manganese priming)
Drug: Sintilimab — Administered intravenously, 200mg on day 3 in a 3-week cycle (day 2 without Manganese priming)
  Other Names: anti-PD-1 antibody; PD-1 inhibitor

SUMMARY:
Ovarian cancer is the most lethal gynecological cancer and the 5th leading cause of cancer death in women. Platinum chemotherapy has been widely adopted as a standard treatment for advanced ovarian cancer, the response rates in patients with relapsed/refractory ovarian cancer is unacceptably low. PD-1 blockade has been developed to a new class of cancer immunotherapy that could restore an adequate immunosurveillance against the neoplasm and enhance T-cell-mediated anticancer immune responses. Manganese has been confirmed to activate antigen-presenting cells and function as mucosal immunoadjuvants in pre-clinical studies. This two-arm, phase I/II study is designed to assess the safety and efficacy of combined therapy of anti-PD-1 antibody and chemotherapy with or without Manganese priming.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically proven relapsed or refractory ovarian cancer (Refractory was defined as a lack of response to or progression during the frontline treatment; relapsed was defined as progression after the frontline treatment), including patients diagnosed with primary carcinoma of fallopian tube or peritoneum carcinoma.
2. Female.
3. ≥ 18 years old.
4. Life expectancy of at least 6 months.
5. Eastern Cooperative Oncology Group performance status 0-2.
6. Radiographic imaging (CT/MRI/PET-CT) indicated recurrence or metastasis; or cancer cells in ascites are positive; or CA125 concentration in the peripheral blood is more than 2 times the upper limit of normal value.
7. Subjects must have received at least two frontline therapies, at least one of which is platinum-containing.
8. Subjects with Anti-PD-1 antibody treatment history are eligible which must be resistance.
9. Adequate organ function.
10. Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study drug.

Exclusion Criteria:

1. Subjects with any autoimmune disease or history of syndrome that requires corticosteroids or immunosuppressive medications.
2. Serious uncontrolled medical disorders or active infections, pulmonary infection especially.
3. Prior organ allograft.
4. Women who are pregnant or breastfeeding.
5. Women with a positive pregnancy test on enrollment or prior to investigational product administration.
6. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
7. Subjects with previous or concurrent other malignancies.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Object response rate (ORR) | 24 months
  ORR is defined as the proportion of subjects who achieved a partial response (PR) or complete response (CR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Number of Subjects with treatment-related adverse events (AEs) | 12 months
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0. AEs were considered to be treatment-related if they had started or worsened within the interval from first study drug administration until the follow-up visit.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 12 months
  DCR is defined as the proportion of subjects who achieved a stable disease (SD), partial response (PR) or complete response (CR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Progression-free survival (PFS) | 12 months
  PFS time was measured from study entry to the first documentation of disease progression or death. Disease progression was determined per the RECIST V1.1.
Overall survival (OS) | 24 months
  OS time was measured from the study entry to the date of death.
Number of participants with laboratory test abnormalities | 12 months
  The laboratory tests of serum cytokines and chemokines will be performed on day 1 and 3 of each cycle, and the abnormality will be determined by the investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China